CLINICAL TRIAL: NCT01881659
Title: Multicentric Study of Cervical Cancer Screening and Triage With Human Papillomavirus (HPV) Testing
Brief Title: Cervical Cancer Screening With Human Papillomavirus Testing
Acronym: ESTAMPA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: IEC 12-27
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: CIN3; CIN2; Cervical Cancer
Keywords: cervical cancer; cancer prevention; cervical screening; HPV testing; triage techniques
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One dry and two liquid cervical samples will be collected at entry. Sample fate will depend on a liquid HPV test. If positive: the dry sample will be used for the E6 protein strip test, the liquid sample for liquid-based cytology and the p16/ki67 test, and 10 aliquots from the second liquid sample will be stored. If negative: the dry sample will be stored for the E6 strip test until the end of the study. Testing will be done based on evidence towards usefulness in primary screening, two aliquots from the first liquid sample will be stored and, the second liquid sample will be discharged. At initial colposcopy, a cervical sample (6 aliquots) and a 10mL blood sample (serum, plasma and buffy-coat) will be collected and stored. All samples will be used for testing of triage techniques.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women attending cervical screening: Women aged 30-64 years who signed informed consent and comply with inclusion and exclusion criteria.
  Interventions: Other: HPV screening

INTERVENTIONS:
Other: HPV screening — Women who signed informed consent will be screened with HPV testing.

SUMMARY:
HPV testing for primary cervical cancer screening of women over 30 years of age is likely to become the standard of care in the near future in many areas of the world. Its high sensitivity can significantly improve the effectiveness of screening programs and its prolonged negative predictive value can allow extension of screening intervals. However, a single HPV test has low positive predictive value and can lead to unnecessary workup and over-treatment and generate unnecessary distress. This multi-centric study will screen 50,000 women with HPV testing and compare several triage approaches that can follow HPV testing in order to make an HPV-based screening programme efficient, affordable and sustainable.

DETAILED DESCRIPTION:
The study will be conducted in several Latin American countries. Currently, the study has started in one site in Colombia and soon another site in Mexico will start. In each participating center, women aged 30-64 years who are attending clinics for cervical screening will be invited to participate in the study. Women who agree to participate and sign the corresponding Institutional Review Board (IRB) approved consent forms will undergo a pelvic examination, and cervical cells for primary screening and triage will be collected. Recruitment specimens will be used for primary screening with an established HPV DNA test (Food and Drug Administration FDA approved). All women who are HPV-positive by the recruitment test will be referred for a standardized colposcopy examination for diagnosis. At the colposcopy visit, but before colposcopy is performed, a risk factor interview will be administered and participants will undergo visual inspection of the cervix with acetic acid (VIA) and collection of additional cervical cells and a blood specimen. The results of VIA will not be disclosed to the colposcopist. During colposcopy, the colposcopists will obtain (2-4) biopsies from any abnormally-appearing areas to ascertain neoplastic outcomes (CIN3+) and to direct treatment as required. All women who attend colposcopy will have a second round of HPV testing approximately 18 months after recruitment and those who are HPV-positive will be referred to colposcopy for final diagnosis. Data management and study supervision will be the responsibility of the International Agency for Research on Cancer (IARC) and the local Principal Investigators, most of whom are experienced HPV researchers.

The combined number of histologically-confirmed diagnoses of CIN3+, including CIN2 lesions positive for p16, (estimated n=500) will be the outcome of primary interest for evaluation of the performance of the various triage modalities. Our initial analyses will focus on comparisons of triage strategies that employ a single method: VIA, conventional/liquid-based cytology, HPV DNA genotyping, HPV RNA detection, detection of E6 proteins of high risk HPV types, or markers of HPV-induced cell-cycle alterations (e.g., p16, ki67, etc). To the extent possible, molecular testing for HPV triage will be carried out on the recruitment specimens to simulate a 'reflex testing' approach wherein screening and triage are done on the same specimen without additional visits. Subsequent analyses will consider various alternative strategies that employ more than one triage methodology; e.g., HPV DNA genotyping followed by cytology. The effectiveness and costs of each alternative strategy will be assessed under various scenarios of feasibility, cost, and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-64 years
* Mentally competent to be able to understand the consent form
* Able to communicate with study staff
* Physically able to have a pelvic exam

Exclusion Criteria:

* Reporting no previous sexual activity
* History of cervical cancer
* Previous treatment for cervical pre-cancer in the last six months
* Hysterectomy
* Plans to move out of the study area in the next 12 months
* Screened for cervical cancer in the last 12 months (depending on local regulations)

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a multicentric study to be carried out in countries across the Latin American region. At each site, a census of all women 28-64 years of age residents of the selected area will be done previously to the start of the study. All women will then be invited using different approaches to the local health centers where screening is to happen.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with histologically confirmed cervical intraepithelial neoplasia grade 3 or cancer (CIN3+), including CIN2 positive for p16, on reviewed histology | Detected after initial HPV screening or at second screening round 18 months since entry
  There will be two HPV screening rounds. Women who test negative for HPV at initial screening will finish their participation. HPV positive women will be: 1) referred to colposcopy, 2) invited for a second HPV screening round if not yet treated, and 3) referred to final colposcopy if HPV positive at second screening. Clinical management will be based on local histology.
  Histology specimens will be externally reviewed by one highly experience international pathologist. If the local and external results are the same, this will become the final histology. If there is disagreement, the specimen will be sent to a third pathologist (be blinded to previous readings). The final diagnosis will then be that agreed by two pathologists (local and either external or both external). Remaining discrepancies will be solved by adjudication at a multi-headed microscope. Worst histology on review will be used to define outcome measures.

SECONDARY OUTCOMES:
Number of participants with histologically confirmed CIN2, CIN3 or cancer (CIN2+) on reviewed histology | Detected after initial HPV screening or at second screening round 18 months since entry
  There will be two HPV screening rounds. Women who test negative for HPV at initial screening will finish their participation. HPV positive women will be: 1) referred to colposcopy, 2) invited for a second HPV screening round if not yet treated, and 3) referred to final colposcopy if HPV positive at second screening. Clinical management will be based on local histology.
  Histology specimens will be externally reviewed by one highly experience international pathologist. If the local and external results are the same, this will become the final histology. If there is disagreement, the specimen will be sent to a third pathologist (be blinded to previous readings). The final diagnosis will then be that agreed by two pathologists (local and either external or both external). Remaining discrepancies will be solved by adjudication at a multi-headed microscope. Worst histology on review will be used to define outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Herrero, MD, PhD, Principal Investigator — International Agency for Research on Cancer (IARC)
Locations (12):
- Argentina (2):
  - Hopsital de Clinicas, Buenos Aires
  - Insituto Malbran - Hospital Posadas, Buenos Aires
- Universidad San Francisco Xavier de Chuquisaca, Sucre, Bolivia
- Colombia (2):
  - National Cancer Institute of Colombia, Bogotá
  - Universidad de Antioquia, Medellín
- Social Security Institute of Costa Rica, San José, Costa Rica
- Universidad Nacional Autonoma de Honduras, Tegucigalpa, Honduras
- Instituto Nacional de Salud Publica de Mexico, Cuernavaca, Morelos, Mexico
- Paraguay (2):
  - Instituto de Investigaciones en Ciencias de la Salud, Universidad Nacional de Asuncion, Asunción
  - Laboratorio Central de Salud Publica, Asunción
- Hospital Santa Rosa, Lima, Peru
- Comision Honoraria de Lucha contra el Cancer, Montevideo, Uruguay

REFERENCES:
- [Derived] Baena A, Picconi MA, Mendoza L, Ferrera A, Mesher D, Lineros J, Brizuela M, Mongelos P, Cabrera Y, Fellner MD, Zambrana O, Garcia L, Hernandez P, Bobadilla ML, Ramon M, Venegas G, Villagra V, Cruz A, Rodriguez G, Teran C, Calderon A, Wiesner C, Herrero R, Almonte M; ESTAMPA study group. Short-term repeat HPV testing for triaging HPV-positive women in cervical cancer screening. Br J Cancer. 2025 Dec;133(12):1844-1853. doi: 10.1038/s41416-025-03193-0. Epub 2025 Oct 3. PMID 41044173
- [Derived] Baena A, Mesher D, Salgado Y, Martinez S, Villalba GR, Amarilla ML, Salgado B, Flores B, Bellido-Fuentes Y, Alvarez-Larraondo M, Valls J, Lora O, Virreira-Prout G, Figueroa J, Turcios E, Soilan AM, Ortega M, Celis M, Gonzalez M, Venegas G, Teran C, Ferrera A, Mendoza L, Kasamatsu E, Murillo R, Wiesner C, Broutet N, Luciani S, Herrero R, Almonte M; ESTAMPA study group. Performance of visual inspection of the cervix with acetic acid (VIA) for triage of HPV screen-positive women: results from the ESTAMPA study. Int J Cancer. 2023 Apr 15;152(8):1581-1592. doi: 10.1002/ijc.34384. Epub 2022 Dec 7. PMID 36451311
- [Derived] Almonte M, Murillo R, Sanchez GI, Gonzalez P, Ferrera A, Picconi MA, Wiesner C, Cruz-Valdez A, Lazcano-Ponce E, Jeronimo J, Ferreccio C, Kasamatsu E, Mendoza L, Rodriguez G, Calderon A, Venegas G, Villagra V, Tatti S, Fleider L, Teran C, Baena A, Hernandez ML, Rol ML, Lucas E, Barbier S, Ramirez AT, Arrossi S, Rodriguez MI, Gonzalez E, Celis M, Martinez S, Salgado Y, Ortega M, Beracochea AV, Perez N, Rodriguez de la Pena M, Ramon M, Hernandez-Nevarez P, Arboleda-Naranjo M, Cabrera Y, Salgado B, Garcia L, Retana MA, Colucci MC, Arias-Stella J, Bellido-Fuentes Y, Bobadilla ML, Olmedo G, Brito-Garcia I, Mendez-Herrera A, Cardinal L, Flores B, Penaranda J, Martinez-Better J, Soilan A, Figueroa J, Caserta B, Sosa C, Moreno A, Mural J, Doimi F, Gimenez D, Rodriguez H, Lora O, Luciani S, Broutet N, Darragh T, Herrero R. Multicentric study of cervical cancer screening with human papillomavirus testing and assessment of triage methods in Latin America: the ESTAMPA screening study protocol. BMJ Open. 2020 May 24;10(5):e035796. doi: 10.1136/bmjopen-2019-035796. PMID 32448795
- [Derived] Robles C, Wiesner C, Martinez S, Salgado Y, Hernandez M, Lucas E, Lineros J, Romero P, Herrero R, Almonte M, Murillo R. Impact of operational factors on HPV positivity rates in an HPV-based screening study in Colombia. Int J Gynaecol Obstet. 2018 Oct;143(1):44-51. doi: 10.1002/ijgo.12574. Epub 2018 Jul 16. PMID 29944728